CLINICAL TRIAL: NCT03922425
Title: Large Scale Implementation of Community Based Mental Health Care for People With Severe and Enduring Mental Ill Health in Europe
Brief Title: Community-based Mental Health Care for People With Severe and Enduring Mental III Health
Acronym: RECOVER-E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The National Center for Public Health and Analyzes, Bulgaria (Other)
Collaborators: Stichting Trimbos-Instituut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01052019
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder; Schizophrenia; Severe Depression
Keywords: Severe mental illnesses
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Depression; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community mental health team (CMHT) (Experimental): CMHTs will be multidisciplinary; that is, staff will be appointed to the CMHTs that include nurses, social workers, psychiatrists, psychologists, and in this project, a peer expert (a person with lived experience of mental health services). All staff within the CMHT will have defined roles and responsibilities that align with the staff functions, roles and linkages detailed in evidence-based service delivery models for community mental health teams. Participant will randomly be assigned to CMHT that will provide outreach mental health care during the project.
  Interventions: Other: Community mental health team
- Standard care (No Intervention)

INTERVENTIONS:
Other: Community mental health team — CMHT will provide home-based treatment inclusive of crisis resolution services and procedures for early recognition of subclinical psychosis and bipolar disorder, and intensive case management. Integrated care (i.e. health and social care interventions) will be provided to all clients. Furthermore, health and social care evidence-based interventions for severe mental illness (SMI) will be employed during home treatment, such as family-based interventions, motivational interviewing, and cognitive behavioural therapies, combined with medication management and identifying employment (paid and non paid options) and support in finding and maintaining this employment, recovery groups and housing opportunities.
  Other Names: CMHT
  Arms: Community mental health team (CMHT)

SUMMARY:
A single-blinded hybrid effectiveness-implementation trial (Type II), that both evaluates the intervention outcomes (clinical and service use outcomes) through patient-randomization in the implementation sites, as well as evaluates the implementation strategy chosen for the intervention and its impact on implementation outcomes (e.g. adoption, fidelity, acceptability and maintenance (continued implementation) of the intervention).

DETAILED DESCRIPTION:
The overall goal of the study is to contribute to improving the level of functioning and quality of life and mental health outcomes for people with severe and enduring mental ill health (SMI) (schizophrenia, bipolar disorder, depression) by adapting and upscaling the implementation of a community-based service delivery model in Montenegro. Effectiveness component of the trial: Multidisciplinary community mental health teams for people with SMI. The intervention condition offers flexible, assertive community treatment (FACT) in the community for people with SMI. FACT can intensify (e.g. provide more intensive treatment in the form of daily home visits, crisis care at home, more intensive evidence-based psycho-social and pharmacological treatments) or provide less intensive treatment depending on client need. It can also provide less intensive care during non-crisis periods, offering routine home treatment where a combination of psychological and pharmacological treatments (e.g. cognitive behavioral therapy, motivational interviewing, family-based interventions) are offered, as well as care processes (reviewing recovery and crisis/treatment plans, and the clients' Wellness Recovery Action Plan), and social care interventions (assistance in obtaining or maintaining employment, looking for reasonable accommodation options). Care offered in this project in the intervention condition will be provided by a multidisciplinary community mental health team (CMHT), consisting of a diverse set of professionals including psychiatrists, psychologists, nurses, and social workers, that deliver integrated medical and social care that are focused on (symptomatic-, functional- and personal-) recovery. CMHTs will provide home-based treatment inclusive of crisis resolution services and procedures for early recognition of sub-clinical psychosis and bipolar disorder, ACT, and intensive case management. Integrated care (i.e. health and social care interventions) will be provided to all clients. Furthermore, health and social care evidence-based interventions for severe mental illnesses will be employed during home treatment, such as family-based interventions, motivational interviewing, and cognitive behavioral therapies, combined with medication management and identifying employment (paid and unpaid options) and support in finding and maintaining this employment, (Wellness Recovery Action Plan (WRAP) recovery groups and housing opportunities. Comparison condition: Usual care Health care settings and their providers randomized to the control condition receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Current service users, with severe and enduring mental disorder,
* Severe Mental Illnesses - bipolar disorder, severe depression, or schizophrenia

Exclusion Criteria:

* Patients who do not consent to their data being collected
* Patients with acute somatic disorders
* Patients who are under the age of 18 at the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in daily functioning | Baseline, 12 months and 18 months
  World Health Organisation Disability Assessment Schedule 2 (WHODAS2) measures health and disability-level of functioning in 6 domains:Cognition, Mobility, Self-care,Getting along, Life activities, Participation in community activities.The instrument is self-reporting; can be administered by a health worker if needed. Answers are distributed into 5 categories:"none","mild","moderate","severe"and"extreme or cannot do". It ends with 3 items where answers are presented as number of days (when difficulties were present). Score on any dimension ranges 0 to 7, results are depicted in a diagram which reflects relation between dimensions(the higher the score, the lower level of difficulties/better functioning) and changes over time

SECONDARY OUTCOMES:
Change in health-related quality of life | Baseline, 12 months and 18 months
  Euro Quality of Life Index (Euro QoL 5-D 3-L). The instrument measures five dimensions: Mobility, Self-care, Daily activities, Pain/Discomfort and Anxiety/ Depression. Each dimension can be rated at three levels: from no problems to major problems. The five dimensions can be summed into a descriptive health state with 11111 representing no problems in any of the five health dimensions and 33333 indicating major problems in any of the five health dimensions. Second part of the instrument is the Visual Analogue Scale to assess health status at baseline, where 0 signifies worst imaginable health state, and 100 signifies best imaginable health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Center "Nikola Shipkovenky", Sofia, Bulgaria

REFERENCES:
- [Derived] Shields-Zeeman L, Smit F, Wijnen B, Roth C, Wensing M, Petrea I; RECOVER-E consortium; Bolinski F, Bajraktarov S, Dedovic J, Keet R, Rojnic Kuzman M, Nakov V, Nica R, Novotni A, Tomcuk A, Djurisic T, Morales G, Rotaru Anghelescu T; RECOVER-E study. Community versus institutionalised care for people with severe mental illness in five countries in Southeast Europe: pooled analysis of five randomised trials. BMJ Glob Health. 2025 Oct 23;10(10):e018594. doi: 10.1136/bmjgh-2024-018594. PMID 41130742
- [Derived] Roth C, Wensing M, Kuzman MR, Bjedov S, Medved S, Istvanovic A, Grbic DS, Simetin IP, Tomcuk A, Dedovic J, Djurisic T, Nica RI, Rotaru T, Novotni A, Bajraktarov S, Milutinovic M, Nakov V, Zarkov Z, Dinolova R, Walters BH, Shields-Zeeman L, Petrea I. Experiences of healthcare staff providing community-based mental healthcare as a multidisciplinary community mental health team in Central and Eastern Europe findings from the RECOVER-E project: an observational intervention study. BMC Psychiatry. 2021 Oct 24;21(1):525. doi: 10.1186/s12888-021-03542-2. PMID 34689733
- [Derived] Wijnen BFM, Smit F, Uhernik AI, Istvanovic A, Dedovic J, Dinolova R, Nica R, Velickovski R, Wensing M, Petrea I, Shields-Zeeman L. Sustainability of Community-Based Specialized Mental Health Services in Five European Countries: Protocol for Five Randomized Controlled Trial-Based Health-Economic Evaluations Embedded in the RECOVER-E Program. JMIR Res Protoc. 2020 Jun 1;9(6):e17454. doi: 10.2196/17454. PMID 32476658
- [Derived] Shields-Zeeman L, Petrea I, Smit F, Walters BH, Dedovic J, Kuzman MR, Nakov V, Nica R, Novotni A, Roth C, Tomcuk A, Wijnen BFM, Wensing M. Towards community-based and recovery-oriented care for severe mental disorders in Southern and Eastern Europe: aims and design of a multi-country implementation and evaluation study (RECOVER-E). Int J Ment Health Syst. 2020 Apr 22;14:30. doi: 10.1186/s13033-020-00361-y. eCollection 2020. PMID 32336984